CLINICAL TRIAL: NCT03809780
Title: Multicenter Phase II Study to Demonstrate Clinical Benefit of Lenalidomide and Dexamethasone in Elderly Unfit Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Study to Demonstrate Clinical Benefit of Lenalidomide and Dexamethasone
Acronym: LENDER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kosin University Gospel Hospital (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Ho Sup Lee, MD, PhD. professor. Division of hematology-Oncology, Kosin University Gospel Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LENDER
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Elderly unfit patients with newly diagnosed multiple myeloma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenalidomide,dexamethasone (Experimental): * High dose for intermediate risk group: lenalidomide 25mg day 1-21 plus dexamethasone 20mg weekly, every 4 weeks
  * Low dose for high risk group: lenalidomide 15mg day 1-21 plus dexamethasone 10mg weekly, every 4 weeks Schedule
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — -high dose: [lenalidomide 25mg day 1-21 plus dexamethasone 20mg weekly] -Low dose: [lenalidomide 15mg day 1-21 plus dexamethasone 10mg weekly]
Drug: Dexamethasone — -high dose: [lenalidomide 25mg day 1-21 plus dexamethasone 20mg weekly] -Low dose: [lenalidomide 15mg day 1-21 plus dexamethasone 10mg weekly]

SUMMARY:
Recent prospective multicenter phase II study assessed the efficacy and tolerability of lower dose lenalidomide (15mg) and dexamethasone (20mg) in frail patients with relapsed or refractory MM. The overall response rate was 71% including complete remission of 15%. Median progression free survival and overall survival were 8.9 and 30.5 months. In addition, grade 3-4 toxicities such as neutropenia, and infections were reduced. This study supported that lower dose lenalidomide may be optimal stating dose for elderly patients with frailty.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignant plasma cell disorder that occurs mainly in older adults. The median age at diagnosis is approximately 70 years, and two-thirds of patients with newly diagnosed MM are older than 65years. As life expectancy increases, the population of older individuals grows. Consequently, the number of patients with MM, especially elderly patients, is expected to increase considerably in the next two decades. Elderly patients may have a variety of comorbidities and reduced physical function at diagnosis, and may be intolerable to standard chemotherapy.

Recent prospective multicenter phase II study assessed the efficacy and tolerability of lower dose lenalidomide (15mg) and dexamethasone (20mg) in frail patients with relapsed or refractory MM[8]. The overall response rate was 71% including complete remission of 15%. Median progression free survival and overall survival were 8.9 and 30.5 months. In addition, grade 3-4 toxicities such as neutropenia, and infections were reduced. This study supported that lower dose lenalidomide may be optimal stating dose for elderly patients with frailty.

Therefore, investigators thought that the use of lower dose of lenalidomide in the frail group is expected to increase the effectiveness as it is used for a long time while reducing toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 70 years unfit and ineligible transplantation in patients with newly diagnosed MM.
2. Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
3. Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
4. Symptomatic MM based on standard CRAB criteria.
5. Patient has measurable disease, defined as follows:

   * any quantifiable serum monoclonal protein value (generally, but not necessarily, ≥ 0.5 g/dL of M-protein) and, where applicable,
   * urine light-chain excretion of >200 mg/24 hours. For patients with oligo or non-secretory MM, it is required that they have
   * Measurable plasmacytoma > 2 cm as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan) or an abnormal free light chain ratio (n.v.: 0.26-1.65). We anticipate that less than 10% of patients admitted to this study will be oligo- or non-secretory MM with free light chains only in order to maximize interpretation of benefit results.
6. The frailty of the patient will be calculated by R-MCI and scoring according to renal function, pulmonary function, activity, frailty, age, and cytogenetics, 0-3 points are low risk (fit) risk (inadequate) and 7 or higher will be classified as high risk (frail). Only inadequate and frail can be included.
7. Patients must meet the following clinical laboratory criteria with 21 days of starting treatment:

   * Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet ≥ 50,000/mm3 (≥ 30,000/mm3 if myeloma involvement in the bone marrow is >50%)
   * Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN.
   * Calculated creatinine clearance ≥ 30mL/min or creatinine < 3mg/dL.
8. Patients who are planned to receive lenalidomide according to license of lenalidomide and must be registered the Risk Management Program(Pregnancy Prevention Program) of each company.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Male patients not agreeing to use an acceptable method for contraception (i.e., condom or abstinence) for the duration of the study.
3. Females of childbearing potential not agreeing to use two acceptable methods for contraception (e.g. a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
4. Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid < to the equivalent of dexamethasone 40 mg/day for 4 days).
5. Any significant medical disease or conditions that, in the investigator's opinion, may interfere with protocol adherence or subject's ability to give informed consent or could place the subject at unacceptable risk.
6. Presence of clinical active infectious hepatitis type B or C, classified into Child-Pugh class C (see Appendix V) and HIV.
7. Presence of acute active infection requiring antibiotics or infiltrative pulmonary disease.
8. Contraindication to any of the required drugs or supportive treatments.
9. prior history of malignancies, other than MM, unless the subject had been free of disease for >= 3 years with the following exceptions: Basal cell CA of skin, Squamous cell CA of skin, CA in situ of cervix and breast, incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)
10. Known allergy to any of the study medications, their analogues, or excipients in the various formulations.
11. Subjects with unstable cardiac disease: MI within 6 months before study participation, NYHA heart failure class III-IV, uncontrolled hypertension/atrial fibrillation,
12. Conditions requiring chronic steroid/immunosuppressive therapy such as RA, MS, lupus, that likely need additional steroid/IS treatment in addition to study treatment
13. Grade >=2 Peripheral neuropathy
14. Subjects who are unwilling or unable to undergo antithrombotic therapy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
2 years Progression Free Survival rates | 2year
  To evaluate the progression free survival rates at 2 years

SECONDARY OUTCOMES:
2 years Event-free survival rates | 2year
  To evaluate the event free survival rates at 2 years
2 years Overall Survival rates | 2year
  To evaluate the overall survival rates at 2 years
Overall response rates | assessed for approximately 2 years after administration
  To evaluated the overall response rates, defined as more than partial response.
Incidence of Treatment-Emergent Adverse Events by CTCAE | assessed for approximately 2 years after administration
  To assess the incidence of lenalidomide plus dexamethasone therapy
Optimal dose in frail patients | through study completion, an average of 1 year
  To assess the optimal dose of lenalidomide for frail patients with newly diagnosed multiple myeloma.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Sup Lee, MD, PhD., Principal Investigator — Kosin University Gospel Hospital
Locations (1):
- Kosin University Gospel Hospital, Busan, Western, South Korea

IPD SHARING:
Plan to Share IPD: Undecided